CLINICAL TRIAL: NCT02922400
Title: Social Cognition Assessment in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Collaborators: University of Texas Southwestern Medical Center (Other); Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STU 042011-021
Record Dates: First submitted 2016-09-29; First posted 2016-10-04 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Cognitive Function 1, Social
Keywords: Autism; Traumatic Brain Injury; Schizophrenia; Virtual-Reality Social Cognition Training
MeSH Terms: conditions — Autistic Disorder; Brain Injuries, Traumatic; Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Social Cognition Assessment and Training (Experimental): Assessment and training program to enhance social function
  Interventions: Behavioral: Social Cognition Assessment and Training

INTERVENTIONS:
Behavioral: Social Cognition Assessment and Training — The study includes an assessment and treatment phase: The assessment phase will test the efficacy and feasibility of a battery of measures evaluating social cognition and behavior. Functional magnetic resonance imaging (fMRI) will also be used to investigate functional differences in regions of the brain associated with social cognition and differences in cognitive progressing. The treatment phase will assess the efficacy and feasibility of a strategy-based social skills treatment using a virtual reality platform.
  Other Names: Virtual Reality Social Cognition Training

SUMMARY:
The primary objective of this study is to determine the efficacy and feasibility of a battery of neuropsychological measures evaluating social cognition and behavior in young adults diagnosed with schizophrenia, autism spectrum disorders, or traumatic brain injury (TBI). It also investigates functional differences in regions of the brain associated with social cognition and differences in cognitive processing. Additionally, this study implements a virtual reality intervention to strengthen social cognition skills.

DETAILED DESCRIPTION:
This purpose of the study is to create a comprehensive social cognitive battery and virtual reality therapy that will be useful in determining and treating social deficits in young adults. With such developments, young adults with social cognition impairment may be provided a way to thoroughly evaluate and treat their deficits.

Participants will be screened for eligibility by research staff. Individuals that have met all enrollment criteria and have provided written consent will be entered into the study. Once written consent has been obtained, participants will enter into the assessment phase of the study, followed by the treatment phase. Both neuropsychological social-cognitive testing and functional magnetic resonance imaging (fMRI) measures will be administered prior and following the treatment phase of the study. The treatment phase will entail use of a virtual-reality platform in which to train and practice social interaction skills. Participants will be reimbursed for the pre- and post- assessment portions only. No compensation will be provided for completing the training.

The first scheduled assessment visits will assess the efficacy and feasibility of a battery of standardized measures as well as measures that are being developed specifically for use with this population, assessing mainly social skills and face processing. The pre-training neuropsychological assessment visit is estimated to take up to 4 hours to complete, however can take longer due to each individual's processing style and social-cognitive abilities. Participants will be scheduled for appointments to conduct both the neuropsychological testing and be given the option to complete an fMRI assessment. The pre-training fMRI assessment visit is estimated to take 1 to 1.5 hours to complete.

Once participants have completed the pre-training assessment, they will enter into the treatment phase of the study and participate in the Virtual Reality Social Cognition Training. Participants will be seen 1-2 times a week for up to six weeks. Session length may range in time from 1 hour to 2 hours each week. Each visit will consist of the participant and clinician engaging in a semi-structured live conversation over a virtual-reality platform. Both the participant and the clinician will talk and interact within the virtual environment through a digital character, an avatar. Each conversation will be set-up, initiated, and conducted by coach and/or confederate clinicians that have been trained to administer the treatment. The confederate clinician will be able to change his/her likeness and voice (through voice modulation software) so as to play the role of the conversation partner with the participant. Live feedback and coaching will be provided by the coach clinician to build social reasoning and thinking skills. Each session will center around a specific social objective (e.g., initiating conversation, conducting a job interview, confronting a friend, going on a blind date) while allowing practicing of specific social strategies. Social strategies will be presented in a hierarchical manner, increasing in complexity throughout the training, to strengthen awareness of and application of social reasoning and thinking skills. Strategies practiced include: 1)recognizing other's social intentions, 2)social response, and 3)self-assertion and social problem solving.

Following completion of the treatment phase, participants will complete post-assessment measures that include neuropsychological social cognitive assessments and an fMRI imaging assessment. The post-neuropsychological assessment visit is estimated to take up to 3 hours to complete where as the post- fMRI visit is estimated to take 1 to 1.5 hours to complete.

ELIGIBILITY:
Inclusion Criteria:

* Current primary diagnosis of schizophrenia, schizoaffective disorder, or autism spectrum disorders as defined by the Diagnostic and Statistical Manual of Mental Disorders, Traumatic Brain Injury (TBI), or healthy control.
* Between the ages of 17 and 40
* TBI must be a close-head injury, at least one year post-injury
* Intelligence Quotient (IQ) at least 80 or above
* Mean Length of Utterance (MLU) must be 4-5 words.

Exclusion Criteria:

* Not fluent in written and oral English
* Clinical status that requires inpatient or day hospital treatment
* Diagnosed with substance dependence within the last three months
* Inability to read self-report instruments
* History of seizures
* Current primary diagnosis of Bipolar Disorder I or II

Ages: 17 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 153 (Actual)
Dates: Start 2006-11; Primary Completion 2016-09 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Brain Activation Change: Social Cognitive Network | Change from Pre-training (prior to treatment) to Post-training (immediately following training)
  To examine activation change in the brain as a result of treatment on fMRI measures to further understand the mechanism and predictors of change in young adults with social impairment.

SECONDARY OUTCOMES:
Change in Neuropsychological Scores: Recognizing Emotion | Change from Pre-training (prior to treatment) to Post-training (immediately following training)
  To examine effects after treatment on the social cognitive skill to recognize emotion
Change in Neuropsychological Scores: Theory of Mind | Change from Pre-training (prior to treatment) to Post-training (immediately following training)
  To examine effects after treatment on the social cognitive skill to have theory of mind, understand other's thought and intentions
Change in Neuropsychological Scores: Social Behavior | Change from Pre-training (prior to treatment) to Post-training (immediately following training)
  To examine effects after treatment on outward social behavior
Change in Neuropsychological Scores: Social Functioning | Change from Pre-training (prior to treatment), to Post-training (immediately following training), and 3-Month follow-up (3 months following completion of training)
  To examine effects after treatment on daily-life social functioning and social engagement

CONTACTS AND LOCATIONS:
Overall Officials: Sandra B Chapman, Ph.D., Principal Investigator — Center for BrainHealth, UT Dallas
Locations (1):
- Center for BrainHealth University of Texas at Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kandalaft MR, Didehbani N, Krawczyk DC, Allen TT, Chapman SB. Virtual reality social cognition training for young adults with high-functioning autism. J Autism Dev Disord. 2013 Jan;43(1):34-44. doi: 10.1007/s10803-012-1544-6. PMID 22570145
- [Result] Didehbani N, Shad MU, Kandalaft MR, Allen TT, Tamminga CA, Krawczyk DC, Chapman SB. Brief report: Insight into illness and social attributional style in Asperger's syndrome. J Autism Dev Disord. 2012 Dec;42(12):2754-60. doi: 10.1007/s10803-012-1532-x. PMID 22527705
- [Result] Didehbani N, Shad MU, Tamminga CA, Kandalaft MR, Allen TT, Chapman SB, Krawczyk DC. Insight and empathy in schizophrenia. Schizophr Res. 2012 Dec;142(1-3):246-7. doi: 10.1016/j.schres.2012.09.010. Epub 2012 Oct 6. No abstract available. PMID 23043874
- [Result] Krawczyk DC, Kandalaft MR, Didehbani N, Allen TT, McClelland MM, Tamminga CA, Chapman SB. An investigation of reasoning by analogy in schizophrenia and autism spectrum disorder. Front Hum Neurosci. 2014 Aug 20;8:517. doi: 10.3389/fnhum.2014.00517. eCollection 2014. PMID 25191240